CLINICAL TRIAL: NCT02821572
Title: Role of Fcgamma Receptors in Immune Thrombocytopenia (ITP)
Acronym: PTI Fc
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: BONNOTTE PARI 2013
Record Dates: First submitted 2016-06-23; First posted 2016-07-01 (Estimated); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Immune Thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- patient
  Interventions: Biological: blood sample; Procedure: spleen sample
- control
  Interventions: Biological: blood sample; Procedure: spleen sample

INTERVENTIONS:
Biological: blood sample
Procedure: spleen sample

SUMMARY:
Immune thrombocytopenia (ITP) is an autoimmune disease characterized by a peripheral destruction of platelets responsible for bleedings.

Monocytes/macrophages play a double role by phagocyting platelets recognized by autoantibodies and by maintaining the autoimmune response via their antigen-presenting cell functions.

Fcgamma receptors (FcγR), that are represented by activating receptors (FcγRI, FcγRIIa, FcγRIII) and an inhibiting one (FcγRIIb), are involved in the regulation of macrophages and have been reported to be dysregulated in autoimmune diseases such as rheumatoid arthritis and systemic lupus erythematous.

The aim of this study is to compare the expression of FcγR in patients with ITP on circulating monocytes and on splenic macrophages.

ELIGIBILITY:
Inclusion Criteria:

ITP group

* Patients who have provided written consent
* Patients over 18 years
* Patients with national health insurance
* Patients with ITP, defined as thrombocytopenia < 100 G/L, after exclusion of infection- or drug-related thrombocytopenia and malignant hemopathy.

Control Group

* Persons who have provided a written consent
* Persons over 18 years
* Persons with national health insurance
* Persons without autoimmune disease

Exclusion Criteria:

* Patients under guardianship
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with ITP Persons without autoimmune disease
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2014-10-02 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
1. The expressions of the activating FcγRs and the inhibiting receptor (FcγRIIb) on monocytes will be compared between ITP patients at diagnosis and controls - physiological parameter | through study completion, an average of 2 years

SECONDARY OUTCOMES:
1. The expressions of the activating FcγRs and the inhibiting receptor (FcγRIIb) on splenic macrophages will be compared between ITP patients and controls. - physiological parameter | through study completion, an average of 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France